CLINICAL TRIAL: NCT03458078
Title: Comparison of the Analgesic Efficacy of Two Adjuvants to Hyperbaric Bupivacaine During Spinal Anaesthesia for Caesarean Section.
Brief Title: Analgesic Efficacy of Two Adjuvants During Spinal Anaesthesia.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre de Maternité de Monastir (Other)
Responsible Party: Principal Investigator, Fethi Jebali, Medical doctor, clinical professor of Anesthesiology and intensive care medecine, Centre de Maternité de Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMMonastir
Record Dates: First submitted 2018-02-15; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Pain, Postoperative
Keywords: Bupivacaine,; Anesthetics; Adjuvants; Analgesics; Peripheral system; Central Nervous; sensory system; Agents; Physiological effects of drugs; opioid; Pain; Postoperative; Signs and Symptoms
MeSH Terms: conditions — Pain, Postoperative; Pain; Signs and Symptoms | interventions — Saline Solution; Sodium Chloride; Magnesium Sulfate; Magnesium; Midazolam; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group C (Placebo Comparator): Control group
  Interventions: Drug: Saline Solution
- Group Mg (Active Comparator): Magnesium sulfate group
  Interventions: Drug: Magnesium Sulfate
- Group MDZ (Active Comparator): Midazolam group
  Interventions: Drug: Midazolam 5 MG/ML Injection

INTERVENTIONS:
Drug: Saline Solution — Spinal injection of 10 mg hyperbaric bupivacaine 0.5% (2 ml) + 100γ morphine (1ml) + 2.5 γ sufentanil (0.5ml) + 1 ml physiological saline.
  Other Names: Saline
  Arms: Group C
Drug: Magnesium Sulfate — Spinal injection of 10 mg hyperbaric Bupivacaine 0.5% (2 ml) + 100γ Morphine (1ml) + 2.5 γ sufentanil (0.5ml) + 100 mg MgSO4 (1 ml).
  Other Names: Magnesium
  Arms: Group Mg
Drug: Midazolam 5 MG/ML Injection — Spinal injection of 10 mg hyperbaric Bupivacaine 0.5% (2 ml) + 100γ Morphine (1ml) + 2.5 γ Sufentanil (0.5ml) + 2mg Midazolam (0.4 + 0.6cc physiological saline (1 ml)).
  Other Names: Midazolam
  Arms: Group MDZ

SUMMARY:
: Pain modulation is very important after operation, particularly for women who undergo caesarean section. A pain-free postoperative period is essential following a caesarean section so new mothers may care for and bond with their neonates. The consequences of the improper pain management which raise the healthcare costs and prolong the recovery process. Intrathecal adjuvants are often administered during this procedure to provide significant analgesia, but they may also have bothersome side effects. Intrathecal midazolam and magnesium sulfate produces effective postoperative analgesia with no significant side effects.

Objectives: This prospective, randomized, double-blind study was designed to compare the analgesic efficacy and safety of intrathecal midazolam vs. Magnesium sulfate vs plain bupivacaine as an adjunct to bupivacaine in pregnancy patients scheduled for elective caesarean section.

DETAILED DESCRIPTION:
The patients were randomly allocated using a computer-generated randomization list to one of three groups that contained 50 parturients each via www.randomization.com.

Group C (control group): 10 mg hyperbaric bupivacaine 0.5% (2 ml) + 100γ morphine (1ml) + 2.5 γ sufentanil (0.5ml) + 1 ml physiological saline.

Group Mg (magnesium sulfate group): 10 mg hyperbaric Bupivacaine 0.5% (2 ml) + 100γ Morphine (1ml) + 2.5 γ sufentanil (0.5ml) + 100 mg MgSO4 (1 ml).

Group MDZ (midazolam group): 10 mg hyperbaric Bupivacaine 0.5% (2 ml) + 100γ Morphine (1ml) + 2.5 γ Sufentanil (0.5ml) + 2mg Midazolam (0.4 + 0.6cc physiological saline (1 ml)).

The parturients as well as the anesthetist who evaluated the protocol did not know the nature of the adjuvant injected in spinal anesthesia. The presented syringe contained one of the two adjuvants or the physiological serum in the same volume and of the same appearance. It was prepared by an anesthesist who was not included in the analysis of the study and was presented anonymously to the anesthetist in charge of the patient. A postoperative monitoring (PO) was performed during the first 24 hours in the intensive care unit by the anesthesist who did not know the nature of the injected adjuvant. All patients were kept nil per os for six hours prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* a mono fetal pregnancy, term> 35 week, planned caesarean section under spinal anesthesia, six-hour fasting, and the American Society of Anesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

* contraindication for intrathecal injection, known allergies to midazolam, other benzodiazepines, magnesium sulfate, caesarean section in extreme urgency, preeclamptic parturient, foetal death in utero, premature delivery (<32SA), anomaly of the placentation, any significant cardiovascular or hepatorenal diseases, a history of seizures or convulsive neurological disease, an altered coagulation profile. Exclusion criteria: failure of spinal anesthesia, conversion into general anesthesia, anesthetic or surgical perioperative incident requiring resuscitation, traumatic puncture, occurrence of serious complication of spinal anesthesia, loss of blindness or randomization of patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
The first requirement for analgesic | 24 hours postoperative
  Postoperatively, the patients were observed for the duration of analgesia using the Visual Analog Scale for Pain (VAS Pain), from 0 - 10 (with 0 being no pain and 10 being the most severe pain imaginable) at H2, H4, H6, H10, H12, H24 at rest and coughing or mobilization until supplementary analgesia was required. The duration of effective analgesia was defined as the time interval between administration of the IT drug to the time of first analgesic request or a VAS ≥ 4. Rescue analgesics were given in the form of a paracetamol injection (1g IV) as well as nefopam (20 mg IV) injection once the VAS was recorded as 4 or more.

SECONDARY OUTCOMES:
The sensory blocks | 24 hours postoperative
  . The assessments of the sensory and motor blocks were taken at the end of each minute until the maximum level of block (T4) was achieved and were assessed using a short, beveled 22-gauge needle and tested at the mid_clavicular line on the chest, trunk, and legs on either side. The duration of the sensory block was defined as the time for regression of the sensory block from the maximum block height to the L-1 dermatome as evaluated by a pinprick.
The motor block | 24 hours postoperative
  The motor block was assessed using the Modified Bromage score (1:Complete block (unable to move feet or knees); 2: Almost complete block (able to move feet only); 3: Partial block (just able to move knees); 4: Detectable weakness of hip flexion while supine (full flexion of knees); 5: No detectable weakness of hip flexion while supine; 6: Able to perform partial knee bend).
Hypotension | 24 hours post operative
  Hypotension was defined as a more than 20% decrease in the systolic blood pressure from the baseline. It was treated with IV fluids and an additional bolus of intravenous (IV) ephedrine (0.1 mg/kg) was repeated at the discretion of the attending anesthesiologist at incremental doses
Bradycardia | 24 hours post operative
  Bradycardia was defined as a decrease in the pulse rate to less than 45 beats per minutes and was treated with an IV injection of 0.5mg atropine sulfate.
Sedation Score | 24 hours post operative
  The sedation scores were recorded using the observer's assessment of the Ramsay scale (Ramsay 1: Anxious, agitated, restless; Ramsay 2: Cooperative, oriented, tranquil; Ramsay 3: Responsive to commands only; Ramsay 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsay 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsay 6: No response to light glabellar tap or loud auditory stimulus).
Maternal satisfaction | 24 hours post operative
  Maternal satisfaction concerning the anesthetic technique was evaluated by the following score:• Excellent = comfort and satisfactory analgesia• Good = average comfort and acceptable analgesia • Poor = significant and lasting discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Rim Cherif, Dr., Study Director — CHU TAHAR SFAR MAHDIA
Locations (2):
- Tunisia (2):
  - Chu Tahar Sfar, Mahdia
  - Centre de Maternité de Monastir, Monastir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakeri H, Pouralborz Y, Askari A, Parkhah M, Hosseinipour A. The adjunctive midazolam or magnesium sulfate to intrathecal bupivacaine analgesic effect in caesarean section: a randomized controlled trial. Biomedical Research. 2017; 28: 3783-3787.